CLINICAL TRIAL: NCT00837993
Title: An Ancillary Study of Patients With Advanced Stage Serous Carcinoma of the Ovary Treated on GOG Protocol 158: A Survival Analysis Based on Reclassification to a Two-tier Grading System
Brief Title: Ancillary Study GOG 158: Survival Analysis Based on Reclassification to a Two-Tier Grading System
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: 2007-0509
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Cancer
Keywords: Advanced Stage Serous Carcinoma of the Ovary; serous ovarian carcinoma; Ovary; GOG Protocol 158; Survival Analysis; Pathology Slides; Two-tier Grading System; Ancillary Study
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survival Analysis: Survival Analysis Based on Reclassification to a Two-tier Grading System: Review of Pathology Slides for Patients participating on Protocol COG 158.

SUMMARY:
Primary Objective:

* To reclassify the histologic grade of the serous ovarian cancer specimens of patients enrolled on Gynecologic Oncology Group (GOG) protocol 158 using a two-tier system.

Secondary Objective:

* To determine the overall and progression-free survival of patients with serous carcinoma of the ovary treated on GOG protocol 158 when reclassified according to tumor grade (low vs. high).

Tertiary Objective:

* To correlate histologic grade with other prognostic factors.

DETAILED DESCRIPTION:
The purpose of this study is to describe the progression-free and overall survival of patients treated on GOG protocol 158 when their tumors are reclassified into a two-tier grading system. Although no universal grading system exists, Malpica et al. have recently published data on a clinically meaningful two-tier grading system for serous ovarian carcinoma (Malpica et al., American Journal of Surgical Pathology, 2004). Tumor grade has been shown to be an important prognostic factor in women with epithelial ovarian cancer, especially in early stage carcinomas. While there is less consensus regarding the prognostic significance of grade in late stage tumors, researchers have noted that patients with low-grade advanced disease may have a longer survival than those with high-grade lesions (Bodurka-Bevers et al., Gynecologic Oncology, 2000).

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled on GOG protocol 158 with a diagnosis of serous carcinoma of the ovary.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients enrolled on GOG protocol 158 with a diagnosis of serous carcinoma of the ovary.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reclassification of histologic grade of the serous ovarian cancer specimens of patients enrolled on Gynecologic Oncology Group (GOG) protocol 158 using a two-tier system. | 2 Years

SECONDARY OUTCOMES:
Overall and Progression-free survival of patients with serous carcinoma of the ovary treated on GOG protocol 158 when reclassified according to tumor grade (low vs. high) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Rose PG, Java JJ, Salani R, Geller MA, Secord AA, Tewari KS, Bender DP, Mutch DG, Friedlander ML, Van Le L, Method MW, Hamilton CA, Lee RB, Wenham RM, Guntupalli SR, Markman M, Muggia FM, Armstrong DK, Bookman MA, Burger RA, Copeland LJ. Nomogram for Predicting Individual Survival After Recurrence of Advanced-Stage, High-Grade Ovarian Carcinoma. Obstet Gynecol. 2019 Feb;133(2):245-254. doi: 10.1097/AOG.0000000000003086. PMID 30633128
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org